CLINICAL TRIAL: NCT05677191
Title: The Usage Of Proximal Femoral Nail Versus Dual Mobility Arthroplasty In Treatment Of Unstable Trochanteric Fractures
Brief Title: PFNA vs Dual Mobility in Treatment of Unstable Trochanteric Fractures
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marcos Hanna Morris, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orthopedic
Record Dates: First submitted 2022-11-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Trochanteric Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Tacrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- proximal femoral nail (Experimental): 20 patient with trochanteric fractures , unstable type will use proximal femoral nail
  Interventions: Device: Proximal Femoral Nail
- Dual Mobility Arthroplasty (Active Comparator): 20 patient with trochanteric fractures , unstable type will use dual mobility arthroplasty
  Interventions: Combination Product: Dual Mobility Arthroplasty

INTERVENTIONS:
Device: Proximal Femoral Nail — open reduction
  Other Names: PFNA
  Arms: proximal femoral nail
Combination Product: Dual Mobility Arthroplasty — Hip Arthroplasty Surgery
  Other Names: THA
  Arms: Dual Mobility Arthroplasty

SUMMARY:
Proximal femoral nail [PFNA] versus dual mobility arthroplasty in treatment of unstable trochanteric fractures

DETAILED DESCRIPTION:
compare clinial outcome between two different procdures either using pfna or arthroplasty in the treatment of unstable trochaneric fractures

ELIGIBILITY:
Inclusion Criteria:

* patients with trochanteric unstable fractures.
* age 60 or above
* recent fracture time within 2 weeks time period
* trochanteric starting point in pfna
* patients medical condition is stable

Exclusion Criteria:

* stable trochanteric fractures
* delayed or neglected fractures
* unstable patients medical conditions
* pirformis fossa starting point in pfna

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip score | Through study completion, an average of 1 year"
  compare between hip score in first group of pfna versus hip score in second group of THA
Operation time | During surgery
  compartive operative time between first group of pfna versus second group of THA